CLINICAL TRIAL: NCT02292589
Title: tDCS in Patients With Mild Traumatic Brain Injury and Persistent Post Concussion Syndrome: Randomized Crossover Trial
Brief Title: Brain Stimulation for Mild Traumatic Brain Injury
Acronym: tDCS/PPCS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: RAHC-001
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Traumatic Brain Injury; Post-Concussion Symptoms
Keywords: Traumatic Brain Injury; Post concussion syndrome; Transcranial Direct Current Stimulation; Neuromodulation
MeSH Terms: conditions — Brain Injuries, Traumatic; Post-Concussion Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Frontal Stimulation (Experimental): Left dorsolateral prefrontal cortex stimulation
  Interventions: Device: Frontal Stimulation
- Temporal Stimulation (Experimental): Left temporal cortex stimulation
  Interventions: Device: Temporal Stimulation
- Sham Stimulation (Experimental): Sham stimulation
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Frontal Stimulation — The patient will receive anodal tDCS on left dorsolateral prefrontal cortex with an intensity of 1.5 mA for 20 minutes.
  Arms: Frontal Stimulation
Device: Temporal Stimulation — The patient will receive anodal tDCS on left temporal cortex with an intensity of 1.5 mA for 20 minutes.
  Arms: Temporal Stimulation
Device: Sham Stimulation — The patient will receive anodal tDCS over the occipital area for 30 seconds only and then it will be turned off without the patient's knowledge.
  Arms: Sham Stimulation

SUMMARY:
The purpose of this study is to determine the early effects of transcranial direct current stimulation (tDCS) in patients with mild traumatic brain injury and persistent post concussion syndrome(PPCS) with cognitive deficits in long term episodic memory and executive function(inhibitory control).

DETAILED DESCRIPTION:
This is a randomized crossover trial of patients with mild TBI (mTBI) sustaining PPCS. It will be recruited twenty adult patients who will receive three sessions of anodal tDCS: left dorsolateral prefrontal cortex, left temporal cortex(with an intensity of 1.5 mA for 20 min) and sham stimulation(intensity of 1.5 mA for 30 seconds only). Sessions will be performed with at least 7 days of interval(wash out period) in a randomized order. Patients who meet the inclusion criteria will be assessed with a neuropsychological evaluation - battery tests include Beck Depression Scale, Hopkins Verbal Learning(HVLT), Stroop test and digit, letters and numbers sequence. A new battery of computerized neuropsychological test will be performed before and immediately after each stimulation(HVLT, Wechsler memory scale, Inhibitory control test(ICT) and block-tapping test.

ELIGIBILITY:
Inclusion Criteria:

* history of mild traumatic brain injury on hospital admission
* subjective complain of memory and executive function
* must be able to sign the Informed Consent Form

Exclusion Criteria:

* under or over age limits
* no specific complain of memory and executive function
* history of major depression(Beck Inventory>35)
* drug addiction
* uncontrolled epilepsy
* presence of any metallic prosthesis implant
* presence of cochlear implant
* not able to sign the Informed Consent Form

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2026-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Evidence of improvement of patient's episodic memory and executive function measured by neuropsychological test | immediately after the stimulation
  HVLT, Wechsler memory scale, Inhibitory control test(ICT) and Block-tapping test.

CONTACTS AND LOCATIONS:
Overall Officials: Robson L Amorim, MD, Principal Investigator — University of Sao Paulo Medical School
Locations (1):
- HC University of Sao Paulo - Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Lesniak M, Polanowska K, Seniow J, Czlonkowska A. Effects of repeated anodal tDCS coupled with cognitive training for patients with severe traumatic brain injury: a pilot randomized controlled trial. J Head Trauma Rehabil. 2014 May-Jun;29(3):E20-9. doi: 10.1097/HTR.0b013e318292a4c2. PMID 23756431
- [Background] Iyer MB, Mattu U, Grafman J, Lomarev M, Sato S, Wassermann EM. Safety and cognitive effect of frontal DC brain polarization in healthy individuals. Neurology. 2005 Mar 8;64(5):872-5. doi: 10.1212/01.WNL.0000152986.07469.E9. PMID 15753425
- [Background] McArthur DL, Chute DJ, Villablanca JP. Moderate and severe traumatic brain injury: epidemiologic, imaging and neuropathologic perspectives. Brain Pathol. 2004 Apr;14(2):185-94. doi: 10.1111/j.1750-3639.2004.tb00052.x. PMID 15193031
- [Background] Bajaj JS, Saeian K, Verber MD, Hischke D, Hoffmann RG, Franco J, Varma RR, Rao SM. Inhibitory control test is a simple method to diagnose minimal hepatic encephalopathy and predict development of overt hepatic encephalopathy. Am J Gastroenterol. 2007 Apr;102(4):754-60. doi: 10.1111/j.1572-0241.2007.01048.x. Epub 2007 Jan 11. PMID 17222319
- [Background] Datta SG, Pillai SV, Rao SL, Kovoor JM, Chandramouli BA. Post-concussion syndrome: Correlation of neuropsychological deficits, structural lesions on magnetic resonance imaging and symptoms. Neurol India. 2009 Sep-Oct;57(5):594-8. doi: 10.4103/0028-3886.57810. PMID 19934558
- [Background] Gorenstein C, Andrade L. Validation of a Portuguese version of the Beck Depression Inventory and the State-Trait Anxiety Inventory in Brazilian subjects. Braz J Med Biol Res. 1996 Apr;29(4):453-7. PMID 8736107
- [Background] King NS. Post-concussion syndrome: clarity amid the controversy? Br J Psychiatry. 2003 Oct;183:276-8. doi: 10.1192/bjp.183.4.276. No abstract available. PMID 14519601
- [Background] Prigatano GP, Gale SD. The current status of postconcussion syndrome. Curr Opin Psychiatry. 2011 May;24(3):243-50. doi: 10.1097/YCO.0b013e328344698b. PMID 21346569
- [Background] Wood RL. Understanding the 'miserable minority': a diasthesis-stress paradigm for post-concussional syndrome. Brain Inj. 2004 Nov;18(11):1135-53. doi: 10.1080/02699050410001675906. PMID 15545210
- [Derived] de Amorim RLO, Brunoni AR, de Oliveira MAF, Zaninotto ALC, Nagumo MM, Guirado VMP, Neville IS, Benute GRG, de Lucia MCS, Paiva WS, de Andrade AF, Teixeira MJ. Transcranial Direct Current Stimulation for Post-Concussion Syndrome: Study Protocol for a Randomized Crossover Trial. Front Neurol. 2017 May 2;8:164. doi: 10.3389/fneur.2017.00164. eCollection 2017. PMID 28512443